CLINICAL TRIAL: NCT02816996
Title: Managing Patient Comfort During Dermatologic Procedures: A Randomized Controlled Trial
Brief Title: Patient Comfort During Dermatologic Procedures
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northwestern University (Other)
Responsible Party: Principal Investigator, Murad Alam, Professor in Dermatology, Otolaryngology-Head and Neck Surgery, and Surgery, Northwestern University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: STU00203158
Record Dates: First submitted 2016-06-27; First posted 2016-06-29 (Estimated); Last update posted 2021-12-06 (Actual); Status verified 2021-12

CONDITIONS: Pain; Anxiety
MeSH Terms: conditions — Pain; Anxiety Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Hand-holding (Experimental): Subjects will be randomized to be in the handholding, stress ball, or control study arms. The randomization will be 1:1:1.
  Interventions: Procedure: Hand-holding
- Stress Ball (Experimental): Subjects will be randomized to be in the handholding, stress ball, or control study arms. The randomization will be 1:1:1.
  Interventions: Procedure: Stress Ball
- Nothing (No Intervention): Subjects will be randomized to be in the handholding, stress ball, or control study arms. The randomization will be 1:1:1.

INTERVENTIONS:
Procedure: Hand-holding — Subject will have their hand held.
  Arms: Hand-holding
Procedure: Stress Ball — Subject will be given a stress ball to hold.
  Arms: Stress Ball

SUMMARY:
The goal of this study is to find the effect of holding a patient's hand on anxiety and pain during dermatologic procedures.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 and older
* Undergoing a dermatologic procedure
* Willing and able to understand and provide informed consent and communicate with the investigator

Exclusion Criteria:

* Subjects who have wound healing problems
* Subjects who are unable to understand the protocol or to give informed consent
* Subjects with self-reported mental illness or other psychological conditions, such as psychotic disorders, mood disorders, anxiety disorders, cognitive disorders, depression with psychotic features, dissociative disorders

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 135 (Actual)
Dates: Start 2017-01-24 (Actual); Primary Completion 2017-04-26 (Actual); Study Completion 2017-04-26 (Actual)

PRIMARY OUTCOMES:
Anxiety | immediately after dermatologic procedure
  Subjects will complete the 6-item State-Trait Anxiety Inventory (STAI)
Pain | immediately after dermatologic procedure
  Subjects will complete a visual analog scale for pain ranging from "no pain at all" to "worst possible pain."

CONTACTS AND LOCATIONS:
Overall Officials: Murad Alam, MD, Principal Investigator — Northwestern University
Locations (1):
- Northwestern Memorial Hospital, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Yanes AF, Weil A, Furlan KC, Poon E, Alam M. Effect of Stress Ball Use or Hand-holding on Anxiety During Skin Cancer Excision: A Randomized Clinical Trial. JAMA Dermatol. 2018 Sep 1;154(9):1045-1049. doi: 10.1001/jamadermatol.2018.1783. PMID 30027283